CLINICAL TRIAL: NCT03505502
Title: Reducing Blood Loss During Cesarean Myomectomy With Intravenous Versus Topical Tranexamic Acid: a Double-blinded Randomized Placebo-controlled Trial
Brief Title: Reducing Blood Loss During Cesarean Myomectomy With Tranexamic Acid
Acronym: TA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/203/2/18
Record Dates: First submitted 2018-04-07; First posted 2018-04-23 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean Myomectomy; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: a double-blinded randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients were randomized to three groups, each compromised of thirty-five patients according to a three-blocked randomization list which was coded (1 or 2 or 3) at 1:1:1 ratio. The three parallel groups were prepared using a Computer-generated randomization system. The allocated groups will be concealed in serially numbered sealed opaque envelopes that will only be opened after recruitment. The patient allocation will be performed prior to the induction of anesthesia by an independent person, who will not otherwise be involved in this study. The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo arm (Placebo Comparator): group receive i/v saline plus irrigation of the myoma bed with normal saline
  Interventions: Drug: IV tranexamic acid
- IV tranexamic acid group (Experimental): group received IV tranexamic 1gm in normal saline
  Interventions: Drug: IV tranexamic acid
- topical tranexamic acid group (Active Comparator): group received topical tranexamic 2gm in normal saline
  Interventions: Drug: IV tranexamic acid

INTERVENTIONS:
Drug: IV tranexamic acid — in IV tranexamic acid group they received 1-gram tranexamic acid (10 ml) in 100 ml saline infusion or placebo (110 normal saline) by slow intravenous injection at an approximate rate of 1 mL per min.In topical tranexamic acid groupA gauze soaked with 2g tranexamic acid (20 ml) diluted in 100 ml of sodium chloride 0.9% or placebo (120ml of sodium chloride 0.9%.) used to compress the myoma bed for 5 minutes. To ensure a sufficiently high concentration, the tranexamic acid was diluted only to a volume sufficient to moisten a large wound surface. 20 ml moisten at least 1500 cm2.
  Other Names: Topical tranexamic acid

SUMMARY:
This study was a double-blinded randomized controlled study conducted at Aswan University, Egypt from January 2018 to January 2020. Study inclusion criteria were women who attended the outpatient obstetric clinic, seeking antenatal care diagnosed with leiomyomas with pregnancy and with myoma staging from (3 to 6) according to FIGO staging. scheduled to undergo cesarean myomectomy (11) Exclusion criteria were: 1-Patients undergone vaginal delivery.2-Patients with a history of thromboembolic disease. 3-Cervical and broad ligament myoma. 4-Myoma FIGO staging

DETAILED DESCRIPTION:
Eligible participants were allocated to one of two groups after induction of anesthesia and immediately prior to the operation and just before skin incision. they received 1-gram tranexamic acid (10 ml) in 100 ml saline infusion or placebo (110 normal salines) by slow intravenous injection at an approximate rate of 1 mL per min. The abdomen was exposed through a midline or Pfannenstiel incision, after skin incision, the subcutaneous fat and abdominal fascia were opened crosswise, and the rectus muscle was opened on the midline. The parietal peritoneum was opened longitudinally to reach the pelvic cavity. Uterus was inspected for a number, location, and shape of myomas and other pelvic organs were inspected for associated pathology. a lower uterine incision will be performed to deliver the baby and Uterine incisions on top of myoma were performed. The incision was performed using monopolar diathermy. Intracapsular enucleation of myomas was performed by gently dissecting between the myoma and the pseudo-capsule. The myoma was grasped by Collins forceps and gently enucleated out.,. Myoma bed was closed by 1 or 2 layers of interrupted vicryl sutures (Vicryl 1-0 polyglactin 910; Egycryl, Taisier CO, Egypt). At the end of the surgery, 1 intraperitoneal suction drain was routinely used in all patients the drains were removed on the second postoperative day unless otherwise indicated. Number and size of myomas were recorded. Myoma size represented the mean size of each myoma. Enucleated myomas were sent to histopathology.

Blood loss estimation Intraoperative blood loss was measured by adding the volume of the contents of the suction bottle and the difference in weight (in grams) between the dry and the soaked operation sheets and towels (1 gram = 1 ml.). Post-operative blood loss was measured through intraperitoneal suction drain which measured every 12 hours and on removing the drain. After that, the total blood loss was calculated by the addition of intraoperative and postoperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* women who attended the outpatient gynecology clinic, seeking treatment for symptomatic leiomyomas and scheduled to undergo abdominal myomectomy with myoma staging from (3 to 6) according to FIGO staging

Exclusion Criteria:

1. Patients undergone vaginal or laparoscopic myomectomy.
2. Patients received preoperative embolization or gonadotrophin releasing hormone analog.
3. Cervical and broad ligament myoma.
4. Patients with cardiac, hepatic, renal or thromboembolic disease
5. patients had an allergy to tranexamic acid).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women who attended the outpatient obstetric clinic, seeking antenatal care diagnosed with leiomyomas with pregnancy and with myoma staging from (3 to 6) according to FIGO staging. scheduled to undergo cesarean myomectomy
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
estimation of intraoperative blood loss (ml). | intraoperative
  Intraoperative blood loss was measured suction bottle and the difference in weight (in grams) between the dry and the soaked operation sheets and towels (1 gram = 1 ml.). Post-operative blood loss was measured through intraperitoneal suction drain which measured every 12 hours and on removing the drain. After that, the total blood loss was calculated by the addition of intraoperative and postoperative blood loss.and vaginal bleeding

SECONDARY OUTCOMES:
need for blood transfusion | 24 hours postoperative
  need for blood transfusion
Hemoglobin concentration | ist 24 hours postoperative
  pre and postoperative hemoglobin estimation
operative time | operative time
  operative time

CONTACTS AND LOCATIONS:
Locations (1):
- AswanUH, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No